CLINICAL TRIAL: NCT03796624
Title: Comparison of Clinical Outcomes After Implantation of MICROPURE (PhysIOL) and PodEye (PhysIOL) Monofocal Intraocular Lenses Into the Two Eyes of the Same Patient
Brief Title: Clinical Outcomes of MICROPURE and PodEye Monofocal Intraocular Lenses
Acronym: PHY1803
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beaver-Visitec International, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHY1803
Record Dates: First submitted 2019-01-04; First posted 2019-01-08 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Cataract; Lens Opacities
Keywords: Intraocular lens; Monofocal; Hydrophobic
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational Device Micropure 1.2.3. (Experimental): Implantation of monofocal intraocular lens (IOL) "Micropure 1.2.3." in one of the eyes of the study subject
  Interventions: Device: Micropure 1.2.3.
- Comparator PODEYE (Active Comparator): Implantation of monofocal intraocular lens (IOL) "PODEYE" in the contralateral eye of the study subject
  Interventions: Device: PODEYE

INTERVENTIONS:
Device: Micropure 1.2.3. — Implantation of intraocular lens (IOL). Name: "MicroPure 1.2.3." It is a monofocal intraocular lens consisting of hydrophobic acrylic material. One IOL per patient will be implanted
  Arms: Investigational Device Micropure 1.2.3.
Device: PODEYE — Implantation of intraocular lens (IOL). Name: "PODEYE" It is a monofocal intraocular lens consisting of hydrophobic acrylic material. The IOL will be implanted in the contralateral eye of the same patient already implanted with Micropure 1.2.3.
  Arms: Comparator PODEYE

SUMMARY:
Prospective, non-randomised, open, controlled, single-center post-market clinical follow study about Micropure 1.2.3. and PODEYE intraocular lenses.

DETAILED DESCRIPTION:
This clinical investigation is a prospective, non-randomised, open, controlled, single-center post-market clinical follow whereby study patients undergoing routine cataract surgery will have implantation of monofocal intraocular lens Micropure 1.2.3. (PhysIOL, Liège, Belgium) in one eye and implantation of monofocal intraocular lens PODEYE (PhysIOL, Liège, Belgium) in the contralateral eye of the same patient.

The study purpose is to obtain clinical data on visual acuity and contrast sensitivity on patients implanted with Micropure 1.2.3. and PODEYE

The devices under investigation (Micropure 1.2.3. and PODEYE) are a monofocal glistening-free hydrophobic acrylic intraocular lenses (IOLs) manufactured by the sponsor of this study PhysIOL sa/nv. The optical properties of the lenses are very comparable. The main difference is the mechanical design of the haptics, that is not expected to have an influence on the clinical outcomes.

The IOLs will be implanted as part of the routine cataract surgery on patients suffering from cataract development.

In total 76 patients will be recruited for this clinical study and receive the implantation of Micropure 1.2.3. and POPDEYE intraocular lenses.

Subjects participating in the trial will attend study visits over a period of 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Cataractous eyes with no comorbidity
* Availability, willingness and sufficient cognitive awareness to comply with examination procedures
* Clear intraocular media other than cataract;
* Signed informed consent

Exclusion Criteria:

* Age of patient < 45 years;
* Irregular astigmatism;
* Regular corneal astigmatism >0.75 dioptres by an automatic keratometer or biometer or >1.0 dioptres if the steep axis of cylinder is between 90° and 120°;
* Difficulty for cooperation (distance from their home, general health condition);
* Previous intraocular or corneal surgery;
* Traumatic cataract;
* Any ocular comorbidity;
* Instability of keratometry or biometry measurements.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2021-06-17 (Actual); Study Completion 2021-06-17 (Actual)

PRIMARY OUTCOMES:
monocular Corrected Distance Visual Acuity (CDVA) | 6 months postoperative
  Statistically non-inferior visual acuity outcomes on monocular Corrected Distance Visual Acuity (CDVA) under photopic light conditions compared to eyes implanted with the comparator PODEYE at the 6 months follow up visit.

SECONDARY OUTCOMES:
Manifested refraction | preoperative, 1 week postoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative
  The manifested refraction is measured by means of a phoropter. The data contains values for sphere, cylinder and axis of cylinder according to ISO 11979-7:2018.
Monocular Uncorrected Distance Visual Acuity (UDVA) under photopic light conditions | preoperative, 1 week postoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative
  UDVA is measured with ETDRS charts placed in 4m distance according to ISO 11979-7:2018. This assessment is performed under photopic light conditions
Monocular Uncorrected Distance Visual Acuity (UDVA) under mesopic light conditions | preoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative
  UDVA is measured with ETDRS charts placed in 4m distance according to ISO 11979-7:2018. This assessment is performed under mesopic light conditions
Monocular Corrected Distance Visual Acuity (CDVA) under photopic light conditions | preoperative, 1 week postoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative
  CDVA is measured with ETDRS charts placed in 4m distance with best aided corrective glasses according to ISO 11979-7:2018. This assessment is performed under photopic light conditions
Monocular Corrected Distance Visual Acuity (CDVA) under mesopic light conditions | preoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative
  CDVA is measured with ETDRS charts placed in 4m distance with best aided corrective glasses according to ISO 11979-7:2018. This assessment is performed under mesopic light conditions
Monocular Contrast Sensitivity under photopic light conditions | 6 months postoperative
  Contrast Sensitivity under photopic light conditions using the standardized contrast sensitivity device CSV-1000 (VectorVision)
Monocular Contrast Sensitivity under mesopic light conditions | 6 months postoperative
  Contrast Sensitivity under mesopic light conditions using the standardized contrast sensitivity device CSV-1000 (VectorVision)
Slitlamp examination - Corneal status | preoperative, 1 week postoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • Corneal status.
Slitlamp examination - Fundus | preoperative, 12 months postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • Fundus.
Slitlamp examination - Signs of inflammation | preoperative, 1 week postoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • Signs of inflammation.
Slitlamp examination - Pupillary block | preoperative, 1 week postoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • Pupillary block.
Slitlamp examination - Retinal detachment | preoperative, 1 week postoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • Retinal detachment.
Slitlamp examination - Status of anterior and posterior capsule | preoperative, 1 week postoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • Status of anterior and posterior capsule.
Slitlamp examination - IOL decentration | preoperative, 1 week postoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • IOL decentration.
Slitlamp examination IOL tilt | preoperative, 1 week postoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • IOL tilt.
Slitlamp examination - IOL discoloration | preoperative, 1 week postoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • IOL discoloration.
Slitlamp examination - IOL opacity | preoperative, 1 week postoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • IOL opacity.

OTHER OUTCOMES:
Intraocular pressure (IOP) measurement | preoperative, 1 week postoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative
  The IOP will be measured with non-contact tonometer as part of the routine follow up examinations
Questionnaire on IOL implantation | peroperative
  A questionnaire will be handed out to the surgeon right after the surgery to document the ease of use and possible issues during IOL implantation. These data will be used to compare the outcomes to different surgery techniques or injectors. The questionnaire is not validated and the outcomes serve only for the sponsor to receive feedback if one or the other IOL is easier to implant.
Keratometry | preoperative
  Keratometric measurements are performed to calculate the required IOL power
Biometry | preoperative
  Biometry measurements are performed to calculate the required IOL power

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Stodůlka, MD, PhD, Principal Investigator — Gemini Eye Clinic
Locations (1):
- GEMINI Eye Clinic, Zlín, Czechia

IPD SHARING:
Plan to Share IPD: No